CLINICAL TRIAL: NCT02569268
Title: Early Vascular Disease Detection System for High Risk Patients in Beijing
Brief Title: Beijing Vascular Disease Patients Evaluation STudy
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Peking University Shougang Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Peking University Health Science Center (Other); Beijing Municipal Science & Technology Commission (Other); Chinese National Natural Science Foundation Commission (Unknown); Ministry of Education, China (Other Government); National Health and Family Planning Commission of the China (Unknown)
Responsible Party: Principal Investigator, Hongyu Wang, Director and Professor of Vascular Medicine, Peking University Shougang Hospital
Other Study IDs: Hongyu Wang
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Vascular Disease
Keywords: Arteriosclerosis; Vascular function; Vascular disease early detection system
MeSH Terms: conditions — Vascular Diseases; Arteriosclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood sample for DNA examination
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- exposure population: No special intervention(s) .
  Interventions: Other: Questionnaires and follow-up

INTERVENTIONS:
Other: Questionnaires and follow-up — Detecting the vascular functional parameters, questionnaire and follow-up: For 2 years or the occurrence of vascular events end time, including cardiovascular events (acute myocardial infarction, angina, coronary reperfusion therapy), stroke, heart failure, peripheral vascular disease.

SUMMARY:
Arteriosclerotic vascular-related diseases have become a serious threat to human health. The prevention and reversal of vascular events has become an important direction of medicine. Early vascular disease detection system includes pulse wave velocity (PWV), carotid intima-media thickness (IMT) and coronary flow velocity reserve (CFVR), flow-mediated vasodilation (FMD), cardio-ankle vascular index (CAVI), ankle-brachial index (ABI), insulin resistance index (HOMA-IR), hypersensitivity C- reactive protein (hs-CRP), plasma homocysteine (Hcy), B-type natriuretic peptide (BNP), uric acid (UA), and so on. However, there is no international and domestic comprehensive study on simple and practical evaluation system by jointing application of these evaluation indexes to detect vascular disease. Combined evaluation function can simultaneously detect and evaluate vascular abnormalities, make up a single indicator shortcoming in clinical applications from multiple levels of vascular structure and function. However, all indicators testing not only cause time consuming, but also increase the burden on patients, resulting unnecessary waste of medical resources. Thus, the present study was to select appropriate indicators and effective joint, and establish the rating system, using the vascular system to predict the incidence of terminal events, and compare this system with the previous scoring system such as FRS (Framingham Risk Score) pros and cons.

DETAILED DESCRIPTION:
This study aimed to establish vascular disease early detection system and scoring systems by comprehensive vascular disease risk factors and vascular function evaluation index. And prevention of vascular-related diseases, high-risk groups through positive lifestyle changes: such as lipid-lowering, smoking cessation, reversing early vascular lesions, to avoid end-stage vascular events.

1. Detection of vascular function indicators include: PWV, IMT, CFVR, FMD, CAVI, ABI, LDL-C, HOMA-IR, hs-CRP, Hcy, BNP, UA and so on.
2. Design the questionnaire: surveying the lifestyle, personal history, family history of the study population.
3. Follow-up:2 years of observation, recording the end time of vascular events, including cardiovascular events (acute myocardial infarction, angina, coronary reperfusion therapy), stroke, heart failure, peripheral vascular disease.
4. Statistics: Complex the factors of vascular disease, screen for an effective indicator to predict cardiovascular events, and based on the weight of the different factors, the establish the rating system, use the system to predict the incidence of vascular events terminal, and compare the system with the previous scoring system such as FRS (Framingham Risk Score).

ELIGIBILITY:
Inclusion Criteria:

1. health subjects with or without history of vascular-related diseases; or
2. hypertension subjects; or
3. diabetes mellitus subjects; or
4. coronary artery disease; or
5. cerebrovascular disease;or
6. hyperlipidemia subjects.

Exclusion Criteria:

1. severe infectious diseases and inflammatory diseases;
2. liver and kidney failure;
3. cancer;
4. immunological diseases;
5. hematological system diseases。

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects such as patient or inpatient patients , aged 45-75 years ,in high-risk vascular events groups ,and from Dongcheng District, Shijingshan Shougang community and Mentougou District.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of vascular diseases-related death | Up to 1 year

SECONDARY OUTCOMES:
Number of acute coronary syndrome | Up to 1 year
  After follow-up and questionnaire, to clear the diagnosis of acute coronary syndrome assessed by guideline or CTCAE v4.0（Grade 3-5).
Number of acute stroke | Up to 1 year
  After follow-up and questionnaire, to clear the diagnosis of acute cerebral infarction and cerebral hemorrhage assessed by guideline.
Number of acute heart failure | Up to 1 year
  After follow-up and questionnaire, to clear the diagnosis of acute heart failure assessed by guideline or CTCAE v4.0（Grade 3-5).
Number of peripheral arteriosclerosis occlusion | Up to 1 year
  After follow-up and questionnaire, to clear the diagnosis of peripheral ischemia by guideline or CTCAE v4.0（Grade 3-5).

REFERENCES:
- [Background] Wang G， He L，Hong T.Reply to letter to the editor: coronary flow velocity reserve was impaired in chronic hyperhomocysteinemia patients：why?Am J Physiol Endocrinol Metab.2011，300：E1177-E1178.
- [Result] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Result] Willum-Hansen T, Staessen JA, Torp-Pedersen C, Rasmussen S, Thijs L, Ibsen H, Jeppesen J. Prognostic value of aortic pulse wave velocity as index of arterial stiffness in the general population. Circulation. 2006 Feb 7;113(5):664-70. doi: 10.1161/CIRCULATIONAHA.105.579342. PMID 16461839
- [Result] Duprez DA, Florea N, Zhong W, Grandits GA, Hawthorne CK, Hoke L, Cohn JN. Vascular and cardiac functional and structural screening to identify risk of future morbid events: preliminary observations. J Am Soc Hypertens. 2011 Sep-Oct;5(5):401-9. doi: 10.1016/j.jash.2011.05.001. Epub 2011 Jun 29. PMID 21719371
- [Result] Hirata K, Kadirvelu A, Di Tullio M, Homma S, Choy AM, Lang CC. Coronary vasomotor function is abnormal in first-degree relatives of patients with type 2 diabetes. Diabetes Care. 2007 Jan;30(1):150-3. doi: 10.2337/dc06-1529. No abstract available. PMID 17192351
- [Result] Ibata J, Sasaki H, Kakimoto T, Matsuno S, Nakatani M, Kobayashi M, Tatsumi K, Nakano Y, Wakasaki H, Furuta H, Nishi M, Nanjo K. Cardio-ankle vascular index measures arterial wall stiffness independent of blood pressure. Diabetes Res Clin Pract. 2008 May;80(2):265-70. doi: 10.1016/j.diabres.2007.12.016. Epub 2008 Feb 1. PMID 18242761
- [Result] Wild SH, Byrne CD, Smith FB, Lee AJ, Fowkes FG. Low ankle-brachial pressure index predicts increased risk of cardiovascular disease independent of the metabolic syndrome and conventional cardiovascular risk factors in the Edinburgh Artery Study. Diabetes Care. 2006 Mar;29(3):637-42. doi: 10.2337/diacare.29.03.06.dc05-1637. PMID 16505519
- [Result] Antoniades C, Antonopoulos AS, Tousoulis D, Marinou K, Stefanadis C. Homocysteine and coronary atherosclerosis: from folate fortification to the recent clinical trials. Eur Heart J. 2009 Jan;30(1):6-15. doi: 10.1093/eurheartj/ehn515. Epub 2008 Nov 23. PMID 19029125
- [Result] He L, Zeng H, Li F, Feng J, Liu S, Liu J, Yu J, Mao J, Hong T, Chen AF, Wang X, Wang G. Homocysteine impairs coronary artery endothelial function by inhibiting tetrahydrobiopterin in patients with hyperhomocysteinemia. Am J Physiol Endocrinol Metab. 2010 Dec;299(6):E1061-5. doi: 10.1152/ajpendo.00367.2010. Epub 2010 Sep 21. PMID 20858749
- [Derived] Liu H, Liu J, Huang W, Zhao H, Zhao N, Wang H. Association between multi-site atherosclerotic plaques and systemic arteriosclerosis: results from the BEST study (Beijing Vascular Disease Patients Evaluation Study). Cardiovasc Ultrasound. 2020 Aug 1;18(1):30. doi: 10.1186/s12947-020-00212-3. PMID 32738905
- [Derived] Liu H, Xie W, Liu J, Zhao H, Wu Y, Wang H. Comparison of vascular-related diseases in their associations with carotid femoral pulse wave velocity: From the Beijing Vascular Disease Patients Evaluation Study (BEST Study). Int J Clin Pract. 2019 Nov;73(11):e13400. doi: 10.1111/ijcp.13400. Epub 2019 Aug 19. PMID 31390128
- [Derived] Lan Y, Liu H, Liu J, Zhao H, Wang H. Gender Difference of the Relationship between Arterial Stiffness and Blood Pressure Variability in Participants in Prehypertension. Int J Hypertens. 2019 Jun 25;2019:7457385. doi: 10.1155/2019/7457385. eCollection 2019. PMID 31341663
- [Derived] Zhao XX, Liu J, Zhao H, Zhou Y, Li L, Wang H. The effect of cardiovascular risk factors on the carotid intima-media thickness in an old-aged cohort with hypertension: a longitudinal evolution with 4-year follow-up of a random clinical trial. Clin Exp Hypertens. 2019;41(1):49-57. doi: 10.1080/10641963.2018.1441860. Epub 2018 Mar 19. PMID 29553852